CLINICAL TRIAL: NCT02495779
Title: Feasibility of Short-Term PrEP Uptake for MSM With Episodic High-Risk for HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Egan (Other)
Collaborators: Fenway Community Health (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, James Egan, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO15060504; 1R34MH104083-01A1 (NIH)
Record Dates: First submitted 2015-06-29; First posted 2015-07-13 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: PrEP; HIV; MSM; Men Having Sex With Men; Episodic PrEP; Adherence; Episodic HIV Risk
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Given emtricitabine/tenofovir for 2-3 weeks. Brief CBT-based counseling to promote PrEP adherence
  Interventions: Drug: emtricitabine/tenofovir; Behavioral: CBT-based counseling

INTERVENTIONS:
Drug: emtricitabine/tenofovir — Short-term episodic use for 2-3 weeks.
  Other Names: Truvada
Behavioral: CBT-based counseling — Brief CBT-based counseling to promote adherence

SUMMARY:
This study is designed to investigate the acceptability, perceived need and uptake of short-term episodic Pre-Exposure Prophylaxis (PrEP) for HIV prevention among men who have sex with men (MSM). The overall objective is to determine the feasibility of a clinic-based Epi-PrEP implementation pilot project for 50 MSM (25/each of the 2 study sites) who report occasional condomless sex and who anticipate a period of high-risk while away from home (e.g. vacation) during the study period.

DETAILED DESCRIPTION:
This proposed study is designed to investigate the acceptability, perceived need and uptake of short-term episodic Pre-Exposure Prophylaxis for HIV prevention among men who have sex with men (MSM). Long-term PrEP may be unnecessary for the many HIV-uninfected men who have episodic contextually defined high-risk periods, particularly when away from their home setting. Alternative dosing strategies, such as short-term fixed-interval episodic PrEP (Epi-PrEP), may be a more realistic, feasible, acceptable, and useful option with high public health impact for the majority of MSM. The overall objective is to determine the feasibility of a clinic-based Epi-PrEP implementation pilot project for 50 MSM (25/each of the 2 study sites) who report occasional condomless sex and who anticipate a period of high-risk while away from home (e.g. vacation) during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as MSM: (1) born male who (2) has sex with men
* Age: 18 or older
* Sexual Risk: has had condomless anal sex with 2 or more men or any transactional sex with a man within the past 12-months.
* Vacation: identified an upcoming period of episodic risk away (i.e. vacation) from their home city that will last at least 7 but not more than 14 days during which they anticipate having at least one high-risk sexual event.
* Able and willing to provide informed consent

Exclusion Criteria:

* HIV positive
* Glomerular filtration rate < 60 mL/min (calculated using the Cockcroft-Gault formula)
* Hepatitis B surface antigen positive
* Symptoms suggestive of acute HIV seroconversion at screening or enrollment
* Have used PrEP or PEP within the previous 3 months
* Currently enrolled in another study involving medications, investigational drug, or medical device
* Has other conditions (based on opinion of investigator or designee) that would preclude informed consent, make the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with study procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Stall, PhD, MPH, Principal Investigator — University of Pittsburgh; Kenneth Mayer, MD, Principal Investigator — Fenway Health
Locations (2):
- United States (2):
  - The Fenway Institute, Boston, Massachusetts
  - Div of Infectious Diseases, University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Egan JE, Ho K, Stall R, Drucker MT, Tappin R, Hendrix CW, Marzinke MA, Safren SA, Mimiaga MJ, Psaros C, Elsesser S, Mayer KH. Feasibility of Short-Term PrEP Uptake for Men Who Have Sex With Men With Episodic Periods of Increased HIV Risk. J Acquir Immune Defic Syndr. 2020 Aug 15;84(5):508-513. doi: 10.1097/QAI.0000000000002382. PMID 32692109

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 54
Completed | 48
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 39
  More than one race | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PrEP Adherence
Description: Biological measure of medication in the blood. Adherence will be measured using plasma analyses. We used the cut off of 4 doses/week to determine protective levels of adherence. The determination of this was drug levels equal to TFV 4.2 ng/mL FTC 4.6 ng/mL.
Time Frame: Blood will be drawn upon within 3 days post-vacation (average 2 weeks after starting PrEP)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 48
Participants | 45

ADVERSE EVENTS:
Time Frame: 4 months
Description: Systematic Assessment of participant reported events at post-trip visit and 3-month follow up.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=48)
HIV seroconverstion (Infections and infestations) | 1 (1) — 1 participant became HIV-infected 2+ months after vacation due to a lapse in insurance to cover ongoing PrEP (move and job change); after 3 months of follow-up there were no other seroconversions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT02495779/Prot_SAP_000.pdf